CLINICAL TRIAL: NCT04075864
Title: Feasibility of a New Model for Exercise Prescription Combined With Behavior Modification in Cystic Fibrosis
Brief Title: Feasibility of a New Model for Exercise Prescription in Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Stefanie Krick MD, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-300003983; UAB (Other: UAB)
Record Dates: First submitted 2019-08-29; First posted 2019-09-03 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Behavior Therapy; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- behavioral intervention to improve physical activity (Experimental): The proposed study is prospective single-arm feasibility clinical trial that will enroll 12 hospitalized patients with CF in accordance with consensus criteria.
  Standard care for an acute CF exacerbation includes i.v. antibiotics and airway clearance therapies for 10-14 days. Routine care following hospitalization is an outpatient CF clinic visit 2-4 weeks after discharge, and then regular follow up every 2-3 months.
  In addition, to standard care in the hospital, study participants will receive a 1) tailored exercise prescription, 2) daily, individual, supervised, aerobic and strength/power training, as well as 3) daily behavioral counseling focused on topics related to long-term adherence to exercise (details below).
  Interventions: Behavioral: Behavioral Counseling and Exercise

INTERVENTIONS:
Behavioral: Behavioral Counseling and Exercise — exercise program combined with behavioral counseling for patients who are hospitalized with a cystic fibrosis exacerbation

SUMMARY:
The purpose of this protocol is to begin an exercise program combined with behavioral counseling for patients who are hospitalized with a cystic fibrosis exacerbation. The exercise program will begin during the hospital stay. Beginning an exercise program during this period of reduced mobility and isolation may be an ideal time to deliver a structured exercise prescription along with a behavioral program to promote long-term adherence to exercise (structured physical activity) . Hospitalized patients have an acute awareness that their lung function is declining and may be more motivated and open to changing their behavior and adding exercise to their treatment regimen.

DETAILED DESCRIPTION:
During the hospitalization (T0 to T1; Figure 1, next page), participants will perform supervised exercise 6 days/wk. On each of these days, there will be a 5-10 min warm up consisting of low intensity execises for lower and upper exermity muscles. The total time per week will be between 2.5 and 3.5 hours.

Three days/wk will consist of aerobic exercise ("frequency"). The various "modes (types)" for this exercise include 1) overground ambulation (including stairs), 2) treadmill ambulation, 3) stationary cycling, or 4) repetitive body-weight exercises (e.g., "jumping jacks"). The "time (duration)" of these sessions will be 20-30 min/day. The "intensity" will be moderate (40-60% of heart rate reserve and/or perceived dyspnea/exertion of 3-5) to vigogous (60-85% of heart rate reserve and/or perceived dyspnea/exertion of 6-8). Participants will be given a HR monitor and specific "target" HR ranges based on their resting HR in standing and their age predicted maximal HR (NOTE: maximal exercise testing will not be performed); they will also be familiarized and instructed in use of the Borg CR10 scale to rate perceived dyspnea/exertion Participants should be able to "talk comfortably" during moderate intensity exercise, while talking should be "somewhat challenging" during vigorous efforts; HR, as well as perceived exertion/dyspnea and "talk test" will be monitored throughout each supervised session by trained personnel.

On alternate days, participants will perform supervised resistance exercise training (3 days/wk; "frequency"). The various "modes (types)" for this exercise include 1) body-weight exercises (e.g., lunges, squats, jumping, situps, pushups) and/or 2) resistance bands and dumbbells; exercises will target upper extremity, trunk/core, and lower extremity muscles (NOTE: specific inspiratory muscle training will not be performed). The "intensity" of these exercises will be at approximately 12-15 repetition max (that is, on the 3rd set of an exercise, the participant should have difficulty performing more than 12-15 quality (good form) repetitions of the exercise. An appropriate number of exercises will be selected such that the exercise "duration (time)" will be 20-30 min/day.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of CF
2. 18 years old or older
3. Current pulmonary exacerbation with planned UAB hospitalization for at least 10 days
4. Willing to participate in a regular, ongoing exercise program
5. Access to broadband internet

Exclusion Criteria:

1. Currently exercising more than 60 min/week
2. Massive hemoptysis or pneumothorax in past 3 months
3. Neuromusculoskeletal impairments that preclude exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
pulmonary function | 1 year
  forced expiratory volume in 1 second

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie Krick, MD, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No